CLINICAL TRIAL: NCT04947553
Title: An Open-Label and Double-Blind, Randomized Withdrawal Study to Assess the Long-term Safety and Efficacy of AXS-05 in Subjects With Dementia of the Alzheimer's Type
Brief Title: A Study to Assess the Long-term Safety and Efficacy of AXS-05 in Subjects With Alzheimer's Disease Agitation
Acronym: ACCORD-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AXS-05-AD-303
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Agitation in Patients With Dementia of the Alzheimer's Type; Alzheimer Disease; Agitation, Psychomotor
Keywords: AD agitation; AXS-05; NMDA receptor antagonist; dextromethorphan; bupropion; Axsome
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-05 (dextromethorphan-bupropion) (Experimental): * Up to 52 weeks in the open-label segment;
  * Up to 24 weeks in the randomized double-blind segment (if applicable)
  Interventions: Drug: AXS-05 (dextromethorphan-bupropion)
- Placebo (Placebo Comparator): Up to 24 weeks in the randomized double-blind segment (if applicable)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-05 (dextromethorphan-bupropion) — AXS-05 tablets, taken twice daily
  Arms: AXS-05 (dextromethorphan-bupropion)
Drug: Placebo — Placebo tablets, taken twice daily
  Arms: Placebo

SUMMARY:
This study will evaluate the long-term safety and efficacy of AXS-05 in subjects with Alzheimer's disease (AD) agitation.

DETAILED DESCRIPTION:
This study is a multi-center trial consisting of an open-label segment of up to 52 weeks, followed by a double-blind, placebo-controlled, randomized withdrawal segment. Subjects participating in the randomized-withdrawal segment will be randomized in a 1:1 ratio either to continue to receive AXS-05 or switch to placebo, for up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Study AXS-05-AD-302 or Study AXS-05-AD-304.
* Caregiver is willing to communicate with site personnel, comply with all required study procedures, and oversee administration and compliance with the subject's study treatment.

Exclusion Criteria:

* Caregiver is unwilling or unable, in the opinion of the investigator, to comply with study instructions.
* Subject is hospitalized in a mental health facility (e.g., psychiatric hospital or ward), living in a nursing home, or living alone.
* Any concurrent medical condition that might interfere with the conduct of the study, confound the interpretation of study results, or endanger the subject's well-being.
* Initiation of a new medication since enrolling in AXS-05-AD-302 or AXS-05-AD-304 which may pose a safety risk when taken concurrently with AXS-05.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 456 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Long-term Safety | up to 76 weeks
  Incidence of treatment-emergent adverse events following dosing with AXS-05
Time to relapse of agitation symptoms | up to 24 weeks

OTHER OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) | up to 76 weeks
  Change from Baseline to last dose in the CMAI

CONTACTS AND LOCATIONS:
Locations (40):
- United States (38):
  - Clinical Research Site, Peoria, Arizona
  - Clinical Research Site, Tempe, Arizona
  - Clinical Research Site, Long Beach, California
  - Clinical Research Site, Santa Ana, California
  - Clinical Research Site, Temecula, California
  - Clinical Research Site, Walnut Creek, California
  - Clinical Research Site, Bonita Springs, Florida
  - Clinical Research Site, Brandon, Florida
  - Clinical Research Site, Coral Springs, Florida
  - Clinical Research Site, Greenacres City, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Hollywood, Florida
  - Clinical Research Site, Kissimmee, Florida
  - Clinical Research Site, Lake City, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Miami Gardens, Florida
  - Clinical Research Site, Miami Lakes, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Pembroke Pines, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Trinity, Florida
  - Clinical Research Site, Columbus, Georgia
  - Clinical Research Site, Wichita, Kansas
  - Clinical Research Site, Braintree, Massachusetts
  - Clinical Research Site, Flint, Michigan
  - Clinical Research Site, Rochester Hills, Michigan
  - Clinical Research Site, Chesterfield, Missouri
  - Clinical Research Site, Toms River, New Jersey
  - Clinical Research Site, Brooklyn, New York
  - Clinical Research Site, New Windsor, New York
  - Clinical Research Site, Staten Island, New York
  - Clinical Research Site, Charlotte, North Carolina
  - Clinical Research Site, Hickory, North Carolina
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Cypress, Texas
  - Clinical Research Site, Mesquite, Texas
  - Clinical Research Site, Sugar Land, Texas
  - Clinical Research Site, Arlington, Virginia
- Clinical Research Site, Kelowna, British Columbia, Canada
- Clinical Research Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com